CLINICAL TRIAL: NCT07198945
Title: Six Versus Twelve Month SurveillAnce Following Resection of Nonpedunculated ColorectaL Polyps 20-50 mm IN Size Without High Grade Dysplasia (HGD)
Brief Title: Six Versus Twelve Month Index Follow-up After Large Colon Polyp Resection
Acronym: STARLING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, John J. Guardiola, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22913
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer; Colon Polyp; Adenoma; Serrated Polyp; Recurrence, Local Neoplasm; Endoscopic Resection
Keywords: Polyp Resection; Colonoscopy; Recurrence; Surveillance Interval; Patient Experience
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Adenoma; Neoplasm Recurrence, Local; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6-month follow-up (Experimental): Patients will be recommended to complete their first surveillance procedure 6 months after the large polyp removal procedure in order to assess whether the polyp grew back.
  Interventions: Procedure: 6-month follow-up
- 12-month follow-up (Experimental): Patients will be recommended to complete their first surveillance procedure 12 months after the large polyp removal procedure in order to assess whether the polyp grew back.
  Interventions: Procedure: 12-month follow-up

INTERVENTIONS:
Procedure: 6-month follow-up — Eligible patients randomized to the 6-month follow-up arm will undergo their first surveillance procedure 6 months after the removal of their large polyp to check for recurrent polyp tissue.
  Arms: 6-month follow-up
Procedure: 12-month follow-up — Eligible patients randomized to the 12-month follow-up arm will undergo their first surveillance procedure 12 months after the removal of their large polyp to check for recurrent polyp tissue.
  Arms: 12-month follow-up

SUMMARY:
The study will compare the use of a 6-month follow-up vs a 12-month follow-up after the removal of a large non-pedunculated polyp 20-50mm in size and without high grade dysplasia.

ELIGIBILITY:
Inclusion Criteria:

Patient Criteria

1. ≥ 18 years of age
2. Ability to provide informed consent
3. Willing and able to complete one electronic survey
4. Presenting for colonoscopy for any indication
5. Ability to understand the requirements of the study and agree to abide by the study restrictions and to return for the required assessments.

   Polyp Criteria
6. Size 20-50 mm as documented with photo containing open snare of known size as comparison.
7. Histology without high grade dysplasia:

   1. Conventional Adenoma: adenoma with or without villous components
   2. Serrated: hyperplastic or sessile serrated lesion

Exclusion Criteria:

Patient Criteria

1. Patients with confirmed diagnosis of inflammatory bowel disease, including Ulcerative Colitis and Crohn's Disease.
2. Patients with a known or suspected diagnosis of any of the following polyposis or non-polyposis syndromes with known genetic mutations:

   * Familial Adenomatous Polyposis Syndrome
   * MUTYH associated Polyposis Syndrome
   * Juvenile Polyposis Syndrome
   * Cowden's Syndrome
   * Peutz-Jeghers Syndrome
   * Hereditary Non-Polyposis Colorectal Cancer Syndrome (HNPCC) or Lynch Syndrome
3. Patients who have high grade dysplasia found in any polyp ≥ 20 mm removed at the index colonoscopy
4. Patients who have any colorectal cancer by histologic diagnosis at index procedure
5. Patients needing a colonoscopy 6 months or sooner for any indication following the index procedure including burden of synchronous disease, inadequate prep to assess for synchronous disease, inadequate prep that precludes resection of index large polyp, or other reason limiting ability to complete full examination of colon at time of resection.
6. ASA ≥ 4 or documented coagulopathy or severe thrombocytopenia (INR ≥ 2 or platelets ≤ 20).
7. Patients who have more than three ≥ 20mm polyps removed during the index colonoscopy
8. Patients with significant acute or chronic medical, neurologic, or illness that, in the judgment of the Principal Investigator, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study.

   Polyp Criteria
9. Polyp located at appendiceal orifice, ileocecal valve, or intradiverticulum
10. Pedunculated or semi-pedunculated polyps (as defined by Paris Classification type Ip or Isp)
11. A polyp that is classified as a traditional serrated adenoma.
12. Polyps with features of invasive cancer
13. Polyps that are not able to be removed with standard endoscopic techniques for any reason
14. Polyps that are incompletely resected endoscopically at index procedure
15. Polyps removed by endoscopic submucosal dissection (ESD) or by full thickness resection device (FTRD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence | 1 day
  Rate of recurrence will be assessed by identification of recurrent polyp tissue at the follow-up procedure.

SECONDARY OUTCOMES:
Time of endoscopic management of recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  The time it takes to treat recurrent polyp at the follow-up procedure
Perceived difficulty of endoscopic treatment of recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  Perceived difficulty of endoscopic treatment of recurrent polyp will be assessed by the endoscopist based at the follow-up procedure on Likert scale 1 - 5 from very difficult to very easy.
Rate of malignancy identified at first surveillance colonoscopy | At first surveillance colonoscopy, typically 6 months to 12 months
  The rate of malignancy measured at the first follow-up colonoscopy
Size of recurrent polyp at first surveillance colonoscopy | At first surveillance colonoscopy, typically 6 months to 12 months
  The size of recurrent polyp tissue as measured by maximum size in millimeters
Number of distinct areas of recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  The number of areas of recurrent polyp tissue identified at the site of the prior large polyp
Rate of high grade dysplasia identified in recurrent polyp | After surveillance colonoscopy, typically 6 months to 12 months
  The rate of high grade dysplasia identified in recurrent polyp tissue.
Need for advanced resection techniques to treat recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  Whether advanced techniques (such as the use of endoscopic submucosal dissection or full thickness resection device) are needed to treat recurrent polyp tissue
Need for surgical intervention to treat recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  Whether surgical intervention is needed to treat recurrent polyp tissue
Types of recurrences at follow-up | At first surveillance colonoscopy, typically 6 months to 12 months
  Description of whether recurrence was visible during the follow-up procedure and confirmed by pathology, visible during the follow-up procedure but not confirmed by pathology, or not visible during the follow-up procedure but confirmed by pathology.
Techniques used to treat recurrent polyp | At first surveillance colonoscopy, typically 6 months to 12 months
  The different techniques that were used to treat the recurrent polyp tissue.
Patient Survey Results | Typically 1 to 14 days after the large polyp removal procedure
  Patient reported experience, including patient's comfort level with prolonged index surveillance, likelihood for returning for follow-up colonoscopy with extended interval, and other factors. This survey is multiple questions, and the responses will be reported on a 5-point Likert scale with 1 being very uncomfortable, not at all important, etc to 5 being very comfortable, very important, etc.
Adverse events that occur after the follow-up procedure | 30 days after first surveillance colonoscopy
  The number of complications for each randomization arm during and after the follow-up procedure
Distance patient travelled to the endoscopy unit | At first surveillance colonoscopy, typically 6 months to 12 months
  Calculation of the distance the patient travelled to the endoscopy unit as a surrogate for carbon impact
Cost of equipment used at the resection site during the follow-up colonoscopy | At first surveillance colonoscopy, typically 6 months to 12 months
  The cost of the equipment that was used at the resection site during the surveillance procedure

CONTACTS AND LOCATIONS:
Overall Officials: John J Guardiola, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared in the future upon request per PI discretion.

REFERENCES:
- [Background] Kaltenbach T, Anderson JC, Burke CA, Dominitz JA, Gupta S, Lieberman D, Robertson DJ, Shaukat A, Syngal S, Rex DK. Endoscopic Removal of Colorectal Lesions-Recommendations by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1095-1129. doi: 10.1053/j.gastro.2019.12.018. Epub 2020 Feb 11. No abstract available. PMID 32122632
- [Background] Gupta S, Lieberman D, Anderson JC, Burke CA, Dominitz JA, Kaltenbach T, Robertson DJ, Shaukat A, Syngal S, Rex DK. Recommendations for Follow-Up After Colonoscopy and Polypectomy: A Consensus Update by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2020 Mar;158(4):1131-1153.e5. doi: 10.1053/j.gastro.2019.10.026. Epub 2020 Feb 7. No abstract available. PMID 32044092
- [Background] El Rahyel A, Abdullah N, Love E, Vemulapalli KC, Rex DK. Recurrence After Endoscopic Mucosal Resection: Early and Late Incidence, Treatment Outcomes, and Outcomes in Non-Overt (Histologic-Only) Recurrence. Gastroenterology. 2021 Feb;160(3):949-951.e2. doi: 10.1053/j.gastro.2020.10.039. Epub 2020 Oct 29. No abstract available. PMID 33130101
- [Background] Tate DJ, Desomer L, Argenziano ME, Mahajan N, Sidhu M, Vosko S, Shahidi N, Lee E, Williams SJ, Burgess NG, Bourke MJ. Treatment of adenoma recurrence after endoscopic mucosal resection. Gut. 2023 Oct;72(10):1875-1886. doi: 10.1136/gutjnl-2023-330300. Epub 2023 Jul 6. PMID 37414440
- [Background] Mohapatra S, Almazan E, Charilaou P, et al. Outcomes of Endoscopic Resection for Colorectal Polyps With High-Grade Dysplasia or Intramucosal Cancer. Techniques and Innovations in Gastrointestinal Endoscopy 2023;25:119-126.
- [Background] Parsa N, Ponugoti P, Broadley H, Garcia J, Rex DK. Risk of cancer in 10 - 19 mm endoscopically detected colorectal lesions. Endoscopy. 2019 May;51(5):452-457. doi: 10.1055/a-0799-9997. Epub 2019 Jan 8. PMID 30620947
- [Background] McWhinney CD, Vemulapalli KC, El Rahyel A, Abdullah N, Rex DK. Adverse events and residual lesion rate after cold endoscopic mucosal resection of serrated lesions >/=10 mm. Gastrointest Endosc. 2021 Mar;93(3):654-659. doi: 10.1016/j.gie.2020.08.032. Epub 2020 Sep 3. PMID 32891621
- [Background] Bobay MC, Lahr RE, Shultz J, Vemulapalli KC, Guardiola JJ, Rex DK. Safety of first surveillance colonoscopy at 12 months after piecemeal EMR of large nonpedunculated colorectal lesions. Gastrointest Endosc. 2024 Nov;100(5):905-913. doi: 10.1016/j.gie.2024.05.008. Epub 2024 May 14. PMID 38750975
- [Background] Lacroute J, Marcantoni J, Petitot S, Weber J, Levy P, Dirrenberger B, Tchoumak I, Baron M, Gibert S, Marguerite S, Huppertz J, Gronier O, Derlon A. The carbon footprint of ambulatory gastrointestinal endoscopy. Endoscopy. 2023 Oct;55(10):918-926. doi: 10.1055/a-2088-4062. Epub 2023 May 8. PMID 37156511
- [Background] Lopez-Munoz P, Martin-Cabezuelo R, Lorenzo-Zuniga V, Vilarino-Feltrer G, Tort-Ausina I, Vidaurre A, Pons Beltran V. Life cycle assessment of routinely used endoscopic instruments and simple intervention to reduce our environmental impact. Gut. 2023 Sep;72(9):1692-1697. doi: 10.1136/gutjnl-2023-329544. Epub 2023 Apr 26. PMID 37185655
- [Background] Belderbos TD, Leenders M, Moons LM, Siersema PD. Local recurrence after endoscopic mucosal resection of nonpedunculated colorectal lesions: systematic review and meta-analysis. Endoscopy. 2014 May;46(5):388-402. doi: 10.1055/s-0034-1364970. Epub 2014 Mar 26. PMID 24671869
- [Background] Pohl H, Rex DK, Barber J, Moyer MT, Elmunzer BJ, Rastogi A, Gordon SR, Zolotarevsky E, Levenick JM, Aslanian HR, Elatrache M, von Renteln D, Wallace MB, Brahmbhatt B, Keswani RN, Kumta NA, Pleskow DK, Smith ZL, Abu Ghanimeh MK, Simmer S, Sanaei O, Mackenzie TA, Piraka C. Cold snare endoscopic resection for large colon polyps: a randomised trial. Gut. 2025 Oct 8;74(11):1804-1813. doi: 10.1136/gutjnl-2025-335075. PMID 40393701